CLINICAL TRIAL: NCT05373381
Title: A Modified Ketogenic, Anti-Inflammatory Diet for Patients With High-Grade Gliomas
Brief Title: The KetoGlioma (Ketogenic Glioma) Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study is on hold indefinitely due to funding issues.
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: KetoGlioma; STUDY00001948 (Other: Tufts Medical Center)
Record Dates: First submitted 2022-04-26; First posted 2022-05-13 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Glioma
Keywords: Glioma; KetoPhyt; High-grade gliomas
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supplemental High Fat Low Carbohydrate (sHFLC) + KetoPhyt (Experimental): Subjects will adhere to the sHFLC + KetoPhyt diet for six 4-week cycles.
  Interventions: Dietary Supplement: Supplemental High Fat Low Carbohydrate (sHFLC) + KetoPhyt

INTERVENTIONS:
Dietary Supplement: Supplemental High Fat Low Carbohydrate (sHFLC) + KetoPhyt — Following a screening period, subjects will adhere to the sHFLC + KetoPhyt diet for six 4-week cycles. Patients will receive dietary advice from a Registered Dietitian (RD) to allow for the design of personalized meal plans maintaining carbohydrates up to 33% of total caloric intake, and be asked to maintain a daily dietary log. To assist patients in understanding, monitoring and controlling their dietary choices to maintain a low carbohydrate diet, they will be trained and receive assistance on the use of an online tool for tracking nutrition [Healthtrac].

SUMMARY:
This research is being conducted to see if patients diagnosed with high grade gliomas can adhere to the supplemented High-Fat Low-Carbohydrate (sHFLC) + KetoPhyt diet, and to see how this diet might affect cancer cells in the bloodstream. This diet is experimental and is not routinely prescribed for patients with high-grade gliomas. The results of this study may be used to support larger studies investigating possible anti-tumor affects of the sHFLC + KetoPhyt diet.

DETAILED DESCRIPTION:
This study is designed to analyze the feasibility of using the sHFLC + KetoPhyt as an anti-cancer agent against glioblastoma multiforme (GBM). While the classic ketogenic diet typically uses a 4:1 ratio of fat to proteins/carbohydrates, the sHFLC + KetoPhyt diet has a maximum 2:1 ratio. This allows increased flexibility in the diet and improved nutritional sufficiency. Preclinical and controlled patient data supports that the sHFLC + KetoPhyt diet is able to decrease blood glucose levels while increasing circulating ketones, two key effects of the ketogenic diet. As caloric restriction is not used in this approach, the investigators hypothesize that patients will be able to have an increased dietary compliance compared to those patients on the very restrictive ketogenic diet, but still achieve a ketotic state.

There is general consensus in the field that the use of the phyto anti-inflammatory diet and exogenous ketone supplementation can all lead to ketosis in a matter of days, and not become what is referred to as ketone adaptative for many weeks to months. Ketosis, with blood levels of the ketone body beta-hydroxy- butarate >0.5 mM, undergoes an adaptive process where different tissues at different times alter the biochemistry of their cellular fuel sources following the switching from a glucose- to fat- and lipid-metabolism. This affects the ability to precisely measure different states of ketosis in the study population over time as the adaptive processes are temporally unique, however previous studies have described the "…adaptation periods necessary… for particular tissue ketone oxidation following sustained nutritional ketosis…" , and these investigators even related this to inflammation-associated cytokine expressions as the investigators propose to measure in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with high-grade gliomas (World Health Organization [WHO] Grade III/IV) with newly diagnosed or recurrent disease
* Ability to understand and willingness to sign an informed consent form prior to any study procedures
* For patients treated with external beam radiation (XRT), interstitial brachytherapy or radiosurgery, an interval of > 4 weeks must have elapsed from completion of XRT to pre-registration.
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2
* Recovered to Common Terminology Criteria for Adverse Events (CTCAE) grade 1 or less toxicity from other agents with exception of alopecia.
* Steroid dosing stable for at least 7 days
* Adequate organ function as defined by the following laboratory values:

  * Absolute neutrophil count (ANC) ≥ 1500/mm3
  * Platelet Count ≥ 100,000/mm3
  * Creatinine ≤ 1.5 mg/dl x upper limit of normal (ULN)
  * Creatinine Clearance ≥ 45 mL/min
  * Total Bilirubin ≤ 1.5 x ULN (except in cases of Gilbert's disease)
  * AST (aspartate aminotransferase)/ ALT (alanine transaminase) ≤ 2.5 x ULN

Exclusion Criteria:

* Concurrent investigational agents or other glioma-directed therapy (chemotherapy, radiation) while on study.
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05-18 (Actual); Primary Completion 2022-05-18 (Actual); Study Completion 2022-05-18 (Actual)

PRIMARY OUTCOMES:
Number of participants not able to adhere the sHFLC + KetoPhyt Diet | From Cycle 1 Day 1 to end of Cycle 6 (Each cycle is 28 days)
  Patients' ability to adhere to the sHFLC + KetoPhyt Diet as defined by the presence of the following:
  1. >75% compliance with taking supplement 2x/day throughout the study period
  2. >75% of days with carbohydrate intake <33%

SECONDARY OUTCOMES:
Change from baseline between the patient's glucose and ketone levels at 24 weeks as assessed by the Glucose/Ketone Index (GKI) | Measured daily from Cycle 1 Day 1 to end of Cycle 6 (Each cycle is 28 days)
  Blood glucose and ketone levels measured at the same time once per day from baseline to 24 weeks via a glucose/ketone monitor and test strips. The Glucose/Ketone Index will be used to monitor patient's glucose and ketone levels.
Change from baseline in pro-inflammatory markers and exosome biomarkers at 24 weeks | At Cycle 1 Day 1 and at Cycle 6 Day 1 (Each cycle is 28 days)
  Comparison of the numbers of EGFrVIII+ exosomes and exosomal microRNAs in each participant's blood measured at baseline (Cycle 1 Day 1) and 24 weeks (Cycle 6).
Change from baseline between the patient's gut microbiome at 24 weeks as assessed by 16s ribosomal sequences. | Measured daily from Cycle 1 Day 1 to end of Cycle 6 (Each cycle is 28 days)
  DNA purified from stool samples (16s ribosomal sequences) will be compared at baseline and 24 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Abdelwahab MG, Fenton KE, Preul MC, Rho JM, Lynch A, Stafford P, Scheck AC. The ketogenic diet is an effective adjuvant to radiation therapy for the treatment of malignant glioma. PLoS One. 2012;7(5):e36197. doi: 10.1371/journal.pone.0036197. Epub 2012 May 1. PMID 22563484
- [Background] Candelario KM, Steindler DA. The role of extracellular vesicles in the progression of neurodegenerative disease and cancer. Trends Mol Med. 2014 Jul;20(7):368-74. doi: 10.1016/j.molmed.2014.04.003. Epub 2014 May 14. PMID 24835084
- [Background] Candelario KM, Balaj L, Zheng T, Skog J, Scheffler B, Breakefield X, Schule B, Steindler DA. Exosome/microvesicle content is altered in leucine-rich repeat kinase 2 mutant induced pluripotent stem cell-derived neural cells. J Comp Neurol. 2020 May;528(7):1203-1215. doi: 10.1002/cne.24819. Epub 2019 Nov 30. PMID 31743443
- [Background] Champ CE, Palmer JD, Volek JS, Werner-Wasik M, Andrews DW, Evans JJ, Glass J, Kim L, Shi W. Targeting metabolism with a ketogenic diet during the treatment of glioblastoma multiforme. J Neurooncol. 2014 Mar;117(1):125-31. doi: 10.1007/s11060-014-1362-0. Epub 2014 Jan 19. PMID 24442482
- [Background] Fadrosh DW, Ma B, Gajer P, Sengamalay N, Ott S, Brotman RM, Ravel J. An improved dual-indexing approach for multiplexed 16S rRNA gene sequencing on the Illumina MiSeq platform. Microbiome. 2014 Feb 24;2(1):6. doi: 10.1186/2049-2618-2-6. PMID 24558975
- [Background] Klein P, Tyrlikova I, Mathews GC. Dietary treatment in adults with refractory epilepsy: a review. Neurology. 2014 Nov 18;83(21):1978-85. doi: 10.1212/WNL.0000000000001004. Epub 2014 Oct 29. PMID 25355830
- [Background] Liu L, Duff K. A technique for serial collection of cerebrospinal fluid from the cisterna magna in mouse. J Vis Exp. 2008 Nov 10;(21):960. doi: 10.3791/960. PMID 19066529
- [Background] Martuscello RT, Vedam-Mai V, McCarthy DJ, Schmoll ME, Jundi MA, Louviere CD, Griffith BG, Skinner CL, Suslov O, Deleyrolle LP, Reynolds BA. A Supplemented High-Fat Low-Carbohydrate Diet for the Treatment of Glioblastoma. Clin Cancer Res. 2016 May 15;22(10):2482-95. doi: 10.1158/1078-0432.CCR-15-0916. Epub 2015 Dec 2. PMID 26631612
- [Background] Meidenbauer JJ, Mukherjee P, Seyfried TN. The glucose ketone index calculator: a simple tool to monitor therapeutic efficacy for metabolic management of brain cancer. Nutr Metab (Lond). 2015 Mar 11;12:12. doi: 10.1186/s12986-015-0009-2. eCollection 2015. PMID 25798181
- [Background] Schwartz K, Chang HT, Nikolai M, Pernicone J, Rhee S, Olson K, Kurniali PC, Hord NG, Noel M. Treatment of glioma patients with ketogenic diets: report of two cases treated with an IRB-approved energy-restricted ketogenic diet protocol and review of the literature. Cancer Metab. 2015 Mar 25;3:3. doi: 10.1186/s40170-015-0129-1. eCollection 2015. PMID 25806103
- [Background] Sherrier M, Li H. The impact of keto-adaptation on exercise performance and the role of metabolic-regulating cytokines. Am J Clin Nutr. 2019 Sep 1;110(3):562-573. doi: 10.1093/ajcn/nqz145. PMID 31347659
- [Background] Siebzehnrubl FA, Reynolds BA, Vescovi A, Steindler DA, Deleyrolle LP. The origins of glioma: E Pluribus Unum? Glia. 2011 Aug;59(8):1135-47. doi: 10.1002/glia.21143. Epub 2011 Feb 23. PMID 21351156
- [Background] Siebzehnrubl FA, Silver DJ, Tugertimur B, Deleyrolle LP, Siebzehnrubl D, Sarkisian MR, Devers KG, Yachnis AT, Kupper MD, Neal D, Nabilsi NH, Kladde MP, Suslov O, Brabletz S, Brabletz T, Reynolds BA, Steindler DA. The ZEB1 pathway links glioblastoma initiation, invasion and chemoresistance. EMBO Mol Med. 2013 Aug;5(8):1196-212. doi: 10.1002/emmm.201302827. Epub 2013 Jul 1. PMID 23818228
- [Background] Skog J, Wurdinger T, van Rijn S, Meijer DH, Gainche L, Sena-Esteves M, Curry WT Jr, Carter BS, Krichevsky AM, Breakefield XO. Glioblastoma microvesicles transport RNA and proteins that promote tumour growth and provide diagnostic biomarkers. Nat Cell Biol. 2008 Dec;10(12):1470-6. doi: 10.1038/ncb1800. Epub 2008 Nov 16. PMID 19011622
- [Background] Strowd RE, Cervenka MC, Henry BJ, Kossoff EH, Hartman AL, Blakeley JO. Glycemic modulation in neuro-oncology: experience and future directions using a modified Atkins diet for high-grade brain tumors. Neurooncol Pract. 2015 Sep;2(3):127-136. doi: 10.1093/nop/npv010. Epub 2015 May 26. PMID 26649186
- [Background] Stupp R, Hegi ME, Mason WP, van den Bent MJ, Taphoorn MJ, Janzer RC, Ludwin SK, Allgeier A, Fisher B, Belanger K, Hau P, Brandes AA, Gijtenbeek J, Marosi C, Vecht CJ, Mokhtari K, Wesseling P, Villa S, Eisenhauer E, Gorlia T, Weller M, Lacombe D, Cairncross JG, Mirimanoff RO; European Organisation for Research and Treatment of Cancer Brain Tumour and Radiation Oncology Groups; National Cancer Institute of Canada Clinical Trials Group. Effects of radiotherapy with concomitant and adjuvant temozolomide versus radiotherapy alone on survival in glioblastoma in a randomised phase III study: 5-year analysis of the EORTC-NCIC trial. Lancet Oncol. 2009 May;10(5):459-66. doi: 10.1016/S1470-2045(09)70025-7. Epub 2009 Mar 9. PMID 19269895
- [Background] Stupp R, Taillibert S, Kanner A, Read W, Steinberg D, Lhermitte B, Toms S, Idbaih A, Ahluwalia MS, Fink K, Di Meco F, Lieberman F, Zhu JJ, Stragliotto G, Tran D, Brem S, Hottinger A, Kirson ED, Lavy-Shahaf G, Weinberg U, Kim CY, Paek SH, Nicholas G, Bruna J, Hirte H, Weller M, Palti Y, Hegi ME, Ram Z. Effect of Tumor-Treating Fields Plus Maintenance Temozolomide vs Maintenance Temozolomide Alone on Survival in Patients With Glioblastoma: A Randomized Clinical Trial. JAMA. 2017 Dec 19;318(23):2306-2316. doi: 10.1001/jama.2017.18718. PMID 29260225
- [Background] Suslov O, Silver DJ, Siebzehnrubl FA, Orjalo A, Ptitsyn A, Steindler DA. Application of an RNA amplification method for reliable single-cell transcriptome analysis. Biotechniques. 2015 Sep 1;59(3):137-48. doi: 10.2144/000114331. eCollection 2015 Sep. PMID 26345506
- [Background] Thery C, Amigorena S, Raposo G, Clayton A. Isolation and characterization of exosomes from cell culture supernatants and biological fluids. Curr Protoc Cell Biol. 2006 Apr;Chapter 3:Unit 3.22. doi: 10.1002/0471143030.cb0322s30. PMID 18228490
- [Background] Truong DT, Franzosa EA, Tickle TL, Scholz M, Weingart G, Pasolli E, Tett A, Huttenhower C, Segata N. MetaPhlAn2 for enhanced metagenomic taxonomic profiling. Nat Methods. 2015 Oct;12(10):902-3. doi: 10.1038/nmeth.3589. No abstract available. PMID 26418763
- [Background] Vlassov AV, Magdaleno S, Setterquist R, Conrad R. Exosomes: current knowledge of their composition, biological functions, and diagnostic and therapeutic potentials. Biochim Biophys Acta. 2012 Jul;1820(7):940-8. doi: 10.1016/j.bbagen.2012.03.017. Epub 2012 Apr 1. PMID 22503788
- [Background] Winter SF, Loebel F, Dietrich J. Role of ketogenic metabolic therapy in malignant glioma: A systematic review. Crit Rev Oncol Hematol. 2017 Apr;112:41-58. doi: 10.1016/j.critrevonc.2017.02.016. Epub 2017 Feb 20. PMID 28325264
- [Background] Woolf EC, Scheck AC. The ketogenic diet for the treatment of malignant glioma. J Lipid Res. 2015 Jan;56(1):5-10. doi: 10.1194/jlr.R046797. Epub 2014 Feb 6. PMID 24503133
- [Background] Zeevi D, Korem T, Zmora N, Israeli D, Rothschild D, Weinberger A, Ben-Yacov O, Lador D, Avnit-Sagi T, Lotan-Pompan M, Suez J, Mahdi JA, Matot E, Malka G, Kosower N, Rein M, Zilberman-Schapira G, Dohnalova L, Pevsner-Fischer M, Bikovsky R, Halpern Z, Elinav E, Segal E. Personalized Nutrition by Prediction of Glycemic Responses. Cell. 2015 Nov 19;163(5):1079-1094. doi: 10.1016/j.cell.2015.11.001. PMID 26590418